CLINICAL TRIAL: NCT00206271
Title: A Randomized Early Intervention Study Comparing the Effect of Stiff Neck Collar, "Act-as-Usual" and Active Mobilisation on the One Year Outcome Following Whiplash Injury.
Brief Title: Comparison of the Effect of Neck Collar, Act-as-Usual, and Active Mobilisation Early After a Whiplash Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Back Research Center, Denmark (Other)
Collaborators: Danish Pain Research Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20000268
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2005-09-21 (Estimated); Status verified 2005-09

CONDITIONS: Whiplash Injury
Keywords: whiplash injuries; neck pain; exercise movement techniques; immobilisation
MeSH Terms: conditions — Whiplash Injuries; Neck Pain

INTERVENTIONS:
Behavioral: neck collar; advice to act-as-usual; active mobilisation

SUMMARY:
Background: Long-lasting pain and disability, known as chronic whiplash-associated disorder (WAD), may develop after forced flexion-extension trauma to the cervical spine. Mechanisms behind WAD are virtually unknown, as are the possible effects of early intervention. This trial was undertaken to compare the effect of three early intervention strategies for the prevention of developing chronic WAD following acute whiplash injury.

Methods: 458 participants were randomised to one of 1) stiff neck collar, 2) advice to act-as-usual, or 3) an active mobilisation regime. Participants were followed for one year and treatment effects were compared in terms of lasting neck pain, headache, disability and sick-leave.

ELIGIBILITY:
Inclusion Criteria:

* Been exposed to rear-end or frontal car collision
* Experienced symptoms within 72 hours
* 18 - 70 years

Exclusion Criteria:

* Could not be enrolled within 10 days of the collision
* Fractures or dislocations of the cervical spine
* Amnesia for the accident
* Unconsciousness in relation to the accident
* Injuries other than the whiplash injury
* Average neck pain during the preceding 6 months exceeding 2 on a box scale 0-10, where 0= no pain and 10= worst possible pain
* Significant pre-existing somatic or psychiatric disease
* Alcohol or drug abuse
* Does not read or understand Danish.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450
Dates: Start 2001-05; Study Completion 2004-10

PRIMARY OUTCOMES:
Neck pain intensity
Headache intensity
Neck disability
Sick leave during the 12 month after inclusion

SECONDARY OUTCOMES:
Medication
Number of non-painful complaints
General health

CONTACTS AND LOCATIONS:
Overall Officials: Tom Bendix, Study Chair — The Back Research Center; Troels S Jensen, Study Chair — Danish Pain Research Center
Locations (2):
- Denmark (2):
  - The Back Research Center, 5750 Ringe
  - Danish Pain Research Center, 8000 Aarhus